CLINICAL TRIAL: NCT00590824
Title: A Pilot Trial of HU14.18-IL2 (EMD273063) in Subjects With Completely Resectable Recurrent Stage III or Stage IV Melanoma
Brief Title: Pilot hu14.18-IL2 in Resectable Recurrent Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2007-0087; CO05601; 2013-1224 (Registry Identifier: Institutional Review Board); NCI-2009-00276 (Registry Identifier: NCI Trial ID); A536755 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison); R01CA032685 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2008-01-11 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Melanoma
Keywords: Melanoma; hu14.18-IL2
MeSH Terms: conditions — Melanoma | interventions — lorukafusp alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Hu14.18-IL2 -->Resection-->Hu14.18-IL2
  Interventions: Drug: hu14.18-IL2
- B (Experimental): Resection -->Hu14.18-IL2-->Hu14.18-IL2
  Interventions: Drug: hu14.18-IL2

INTERVENTIONS:
Drug: hu14.18-IL2 — 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course followed by surgery and up to 2 additional courses of hu14.18-IL2
  Arms: A
Drug: hu14.18-IL2 — Surgery followed by 3 courses of 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course
  Arms: B

SUMMARY:
Evaluate the antitumor activity of hu14.18-IL2 in the minimal residual disease setting. Evaluate the time to recurrence and overall survival of patients treated with hu14.18-IL2.

ELIGIBILITY:
Inclusion criteria

1. Subjects must have recurrent stage III (i.e., recurrent regional metastasis), or stage IV (i.e., any distant metastasis) melanoma for which surgical resection would be clinically recommended, with biopsy proven (current or previous) Stage III or Stage IV disease. Any biopsies obtained to demonstrate recurrent regional metastasis or distant metastasis must be considered clinically appropriate for clinical management and must not be performed solely for meeting eligibility criteria. In addition, subjects must have disease that has not yet been completely excised.
2. Patients must have disease which involves 3 or fewer sites. A nodal basin recurrence will be scored as one site, even if multiple nodes are positive. "Clustered" subcutaneous and/or cutaneous lesions that can be removed in a single surgical excision will be scored as one site, even if multiple subcutaneous and/or cutaneous lesions are present.
3. The subjects' disease is determined to be completely resectable with uninvolved margins using standard surgical guidelines based on physical exam and radiographic imaging (MRI or CT of the head, and CT or MRI of the chest, abdomen and pelvis).
4. Subjects must have one of the following: a) Stage III melanoma with recurrence after prior surgery, with or without subsequent adjuvant systemic (standard or experimental) and/or radiotherapy management Or b) Stage IV melanoma (cutaneous, ocular, mucosal, or unknown primary)
5. Subjects must be 18 years old or older OR if they are 15 years old or greater, considered to be mature minors, able to give adult informed consent (with parental co-signature), meet all other eligibility criteria, and also weigh at least 45 kg.. Subjects must weigh at least 45 kg in order to safely provide sufficient blood for monitoring studies (see section 7.7 for details).
6. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Subjects must have adequate bone marrow, liver, and renal function.
8. Subjects with one or more of the following cardiac risk factors must complete a stress radionuclide scan with no evidence of myocardial ischemia or heart failure: (a) a history of cardiac disease, (b) age greater than 65 years old, (c) any clinically significant abnormality found on ECG (required at baseline), or (d) significant risk factors for coronary artery disease (history of significant dyslipidemia; any treatment for dyslipidemia; or two first degree relatives with a documented myocardial infarction prior to age 55).
9. Subjects with significant history of pulmonary disease, shortness of breath at rest, or known Chronic Obstructive Pulmonary Disease (COPD) must have pulmonary function tests within 35% of normal age-predicted values.
10. Subjects must be willing and able to provide informed written consent prior to any study-related procedures.
11. Subjects must have no immediate requirements for palliative chemotherapy, palliative radiotherapy, or palliative hormonal therapy.
12. Subjects must be willing and able to discontinue antihypertensive medications if advised to do so for days of hu14.18-IL2 infusion.
13. Subjects must have slides available from stage III or stage IV melanoma. Paraffin blocks are preferable, but at a minimum, slides documenting melanoma by biopsy (including fine needle cytology) must be available for pathology review, and potential restaining/staining (see Section 7.4, Surgical Pathology Guidelines). Prior histologic demonstration of metastatic melanoma (either stage III or Stage IV) may be utilized if a repeat biopsy is not clinically needed to to establish eligibility.

Exclusion criteria

1. Subjects are ineligible if they have received monoclonal antibodies (mAb) during biologic therapy, tumor imaging, purging of autologous marrow/stem cells for re-infusion or for any other reason unless serological testing is performed. If the absence of detectable antibody (over background) to hu14.18 is documented, the subject is eligible for the study.
2. Subjects treated with IL2 in the past that developed intolerable (Grade 4) IL2-related side effects are not eligible.
3. Subjects who have received any (standard or experimental) systemic therapy for stage IV disease are not eligible.
4. Women of childbearing potential will be excluded if they are pregnant, nursing, or not using effective contraception during the treatment period.
5. Subjects with symptoms of ischemic cardiac disease, congestive heart failure, myocardial infarct within the immediate preceding 6 months and/or uncontrolled cardiac rhythm disturbance are ineligible.
6. Subjects with significant psychiatric disabilities or seizure disorders are ineligible.
7. Subjects who have had major surgery within the past 3 weeks are ineligible.
8. Subjects with clinically detectable pleural effusions or ascites are ineligible.
9. Subjects with organ allografts are ineligible.
10. Subjects who require or are likely to require corticosteroid or other immunosuppressive drugs or have used them within 2 weeks of registration are ineligible.
11. Subjects with significant intercurrent illnesses are ineligible.
12. Subjects with active infections or active peptic ulcer unless these conditions are corrected or controlled are ineligible.
13. Subjects with brain metastases, whether active or inactive, are ineligible. A head MRI or head CT scan will be required at baseline to rule out silent metastases.
14. Subjects with active second malignancy other than non-melanoma skin cancer are ineligible. Patients will be considered eligible if they have been continuously disease free for > 5 years prior to the time of enrollment.
15. Subjects who are infected with human immunodeficiency virus (HIV), hepatitis B surface antigen (HBs Ag) carrier state or with clinical evidence of hepatitis are ineligible. Treatment may be initiated before laboratory confirmation of HIV and HBs Ag negativity, but will be stopped if results are positive.
16. Subjects with a clinically significant neurologic deficit or objective peripheral neuropathy (Grade > 2) are ineligible.
17. Subjects with a known hypersensitivity to the study drug, Tween-80® or to human immunoglobulin are ineligible.
18. Patients with a known history of diabetes mellitus that has required systemic therapy within the past 3 months (either oral hypoglycemic agents or insulin) will be excluded, as treatment with hu14.18-IL2 may alter blood glucose levels.
19. Subjects with a legal incapacity or limited legal capacity are ineligible.
20. Subjects with bone metastases are ineligible.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Sondel, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Mark R Albertini, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Albertini MR, Yang RK, Ranheim EA, Hank JA, Zuleger CL, Weber S, Neuman H, Hartig G, Weigel T, Mahvi D, Henry MB, Quale R, McFarland T, Gan J, Carmichael L, Kim K, Loibner H, Gillies SD, Sondel PM. Pilot trial of the hu14.18-IL2 immunocytokine in patients with completely resectable recurrent stage III or stage IV melanoma. Cancer Immunol Immunother. 2018 Oct;67(10):1647-1658. doi: 10.1007/s00262-018-2223-z. Epub 2018 Aug 3. PMID 30073390
- [Derived] Yang RK, Kuznetsov IB, Ranheim EA, Wei JS, Sindiri S, Gryder BE, Gangalapudi V, Song YK, Patel V, Hank JA, Zuleger C, Erbe AK, Morris ZS, Quale R, Kim K, Albertini MR, Khan J, Sondel PM. Outcome-Related Signatures Identified by Whole Transcriptome Sequencing of Resectable Stage III/IV Melanoma Evaluated after Starting Hu14.18-IL2. Clin Cancer Res. 2020 Jul 1;26(13):3296-3306. doi: 10.1158/1078-0432.CCR-19-3294. Epub 2020 Mar 9. PMID 32152202
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol amended to drop cilengitide groups (C and D), proceed with enrollment and randomization into hu14.18- IL2 groups.
Groups:
- Group A: Hu14.18-IL2 -->Resection-->Hu14.18-IL2
  hu14.18-IL2: 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course followed by surgery and up to 2 additional courses of hu14.18-IL2
- Group B: Resection -->Hu14.18-IL2-->Hu14.18-IL2
  hu14.18-IL2: Surgery followed by 3 courses of 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course
- Group C: Cilengitide +Hu14.18-IL2-->Resection-->Cilengitide+Hu14.18-IL2
  [This Arm was suspended and subsequently removed from the study design via protocol amendment due to toxicity]
- Group D: Cilengitide-->Resection-->Cilengitide + Hu14.18-IL2
  [This Arm was suspended and subsequently removed from the study design via protocol amendment due to toxicity]
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 11 | 9 | 2 | 1
Completed | 11 | 7 | 1 | 0
Not Completed | 0 | 2 | 1 | 1
Not completed — Disease could not be resected | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Groups C and D were suspended due to toxicity and removed from the study design in a subsequent protocol amendment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 11 | 9 | 2 | 1 | 23
Age, Continuous [Median (Full Range); unit: years] | 46 [21 to 65] | 52 [38 to 69] | 56 [51 to 61] | 67 [67 to 67] | 47 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 0 | 8
  Male | 6 | 7 | 1 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 2 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 2 | 1 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 2 | 1 | 23
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) - criteria are used by doctors and researchers to assess how a patient's disease is progressing on a scale of 0-5 where 0 (Fully active, able to carry on all pre-disease performance without restriction),1 (Restricted in physically strenuous activity but ambulatory), to 5 (Death).
  Participants
    0 | 9 | 7 | 2 | 1 | 19
    1 | 2 | 2 | 0 | 0 | 4
Disease Extent [Count of Participants; unit: Participants]
  Extensive | 4 | 2 | 1 | 0 | 7
  Non-extensive | 7 | 7 | 1 | 1 | 16
Disease Stage [Count of Participants; unit: Participants] — Disease stage indicates the amount the disease has spread (Stage 0-IV). Stage III has spread regionally, is defined by the level of lymph node involvement and has no evidence of metastasis. Stage IV indicates metastasis beyond the original site.
  Participants
    III | 7 | 6 | 0 | 1 | 14
    IV | 4 | 3 | 2 | 0 | 9
Histology [Count of Participants; unit: Participants]
  Cutaneous melanoma | 10 | 8 | 2 | 1 | 21
  Unknown melanoma primary | 1 | 0 | 0 | 0 | 1
  Subungual melanoma | 0 | 1 | 0 | 0 | 1
Prior Therapy [Number; unit: participants]
  Granulocyte-macrophage colony stimulating factor | 1 | 0 | 0 | 0 | 1
  Chemotherapy multiple agent | 0 | 1 | 0 | 0 | 1
  Interferon alpha-2b | 7 | 5 | 1 | 1 | 14
  No prior therapy | 1 | 0 | 0 | 0 | 1
  Radiation therapy | 1 | 2 | 0 | 0 | 3
  Surgery | 10 | 9 | 2 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Ganglioside Expressed by Tumor Cells (GD2)
Description: Histological analysis of anti-tumor activity is a primary endpoint. This is measured after surgical resection via staining to indicate GD2 expression. The GD2 results were summarized in terms of positive (GD2 expression high or low/moderate) and negative (GD2 expression undetectable).
Time Frame: up to 1 week
Population: There were 12 participants with evaluable tumor samples for GD2 analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 6
Participants
  Positive GD2 | 3 | 3
  Negative GD2 | 3 | 3

2. Primary Outcome: Recurrence Free Survival (RFS)
Description: RFS was defined as the number of days from the day of evaluation following course 2 of immunocytokine treatment to the day the subject experienced an event of recurrence or death, whichever occurred first. Participants who did not experience an event of recurrence or death at the time of analysis were censored at the date of the last evaluation for recurrence.
Time Frame: up to 24 months
Population: Two patients in Group B were not treated with adjuvant hu14.18-IL2. Subsequently these two patients were excluded from the RFS analysis. There was no intent in the protocol to compare RFS between Groups A and B.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A and B: Hu14.18-IL2 ->Hu14.18-IL2
  [All participants received same treatment]
  hu14.18-IL2: 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course followed by up to 2 additional courses of hu14.18-IL2
Arm/Group | Group A and B
Number analyzed (Participants) | 18
months | 5.73 [1.80 to NA] — the value is infinity (reported as INF)

3. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the number of days from randomization to the date of the participant's death. Participants who did not experience an event of death at the time of analysis were censored at the date of the last follow-up.
Time Frame: up to 24 months
Population: There was no intent in the protocol to compare OS between Groups A and B.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A and B: Hu14.18-IL2 -->Hu14.18-IL2
  [All participants received the same treatment]
  hu14.18-IL2: 6 mg/m2 hu14.18-IL2 administered via IV on days 1, 2, and 3 of a 28-day course followed by up to 2 additional courses of hu14.18-IL2
Arm/Group | Group A and B
Number analyzed (Participants) | 20
months | 61.57 [13.67 to NA] — the value is infinity (reported as INF)

4. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP measured at baseline, cycle 1 day 3, and cycle 2 day 1.
Time Frame: up to 29 days
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 7
mg/dL
  baseline | 0 [0 to 9] | 0 [0 to 1]
  cycle 1 day 3 | 9 [7 to 14] | 11 [6 to 13]
  cycle 2 day 1 | 0 [0 to 7] | 0 [0 to 4]

5. Secondary Outcome: Lymphocyte Count
Description: Lymphocyte count measured at baseline, cycle 1 day 3, cycle 1 day 8, and cycle 2 day 1
Time Frame: up to 29 days
Measure: Median (Full Range); unit: number of lymphocytes
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 7
number of lymphocytes
  baseline | 1750 [1090 to 2430] | 1440 [960 to 2300]
  cycle 1 day 3 | 200 [62 to 460] | 250 [170 to 270]
  cycle 1 day 8 | 4910 [2610 to 6954] | 3900 [2420 to 4470]
  cycle 2 day 1 | 3160 [1790 to 4110] | 2100 [1730 to 3080]

6. Secondary Outcome: Anti-Idiotypic Antibodies
Description: Detection of anti-idiotypic will be performed on participants' serum obtained approximately 10 minutes prior to initiation of treatment, and serum samples on Days 3, 4, 8, and 29/1 of 3 cycles.
Time Frame: up to 12 weeks
Population: Based on data collected from prior trials and analyzed during the time of this trial, the day 3 sample (obtained during hu14.18-IL2 administration) was potentially "masked" by the infusion of the immunocytokine. Anti-immunocytokine antibodies were not typically generated during the initial 5 days when infusions were given on days 1-3.
Measure: Mean (Standard Error); unit: Optical Density (OD)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 7
Optical Density (OD)
  Cycle 1 Day 1 pre-treatment | 0.2 (0.09) | 0.2 (0.12)
  Cycle 1 Day 4 | 0.4 (0.11) | 0.8 (0.33)
  Cycle 1 Day 8 | 1.5 (0.23) | 1.7 (0.42)
  End Cycle 1 | 0.6 (0.24) | 0.6 (0.18)
  Cycle 2 Day 1 pre-treatment | 0.4 (0.11) | 0.5 (0.13)
  Cycle 2 Day 4 | 0.4 (0.16) | 0.5 (0.17)
  Cycle 2 Day 8 | 1.5 (0.31) | 1.4 (0.23)
  End Cycle 2 | 0.9 (0.24) | 0.6 (0.16)
  Cycle 3 Day 1 pre-treatment | 0.9 (0.28) | 0.5 (0.14)
  Cycle 3 Day 4 | 0.4 (0.09) | 0.6 (0.16)
  Cycle 3 Day 8 | 1.0 (0.30) | 1.2 (0.28)
  End Cycle 3 | 0.7 (0.27) | 0.5 (0.12)

7. Secondary Outcome: Anti-Fc-IL2 Antibodies
Description: Detection of anti-FcIL2 will be performed on participants' serum obtained approximately 10 minutes prior to initiation of treatment, and serum samples on Days 3, 4, 8, and 29/1, for 3 cycles
Time Frame: up to 12 weeks
Population: The investigators determined in real time that the evaluation of anti-Fc-Il2 antibodies was not an appropriate biomarker for this study. The patient generated "anti-drug antibody," specific for the Fc-IL2 component of the immunocytokine is detected in the standard "anti-idiotypic" bridge assay (reported in Outcome Measure 6).
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: In Vitro Soluble Interleukin-2 (IL2) Receptor Alpha Levels
Description: Soluble IL2 receptor α levels will be performed on participants approximately 10 minutes prior to initiation of treatment, and serum samples on Days 3, 4, 8, and 29/1.
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 7
ng/ml
  10 min prior to initiation of Cycle 1 treatment | 1293.0 (150.1) | 1229.7 (260.8)
  Cycle 1 Day 3 | 6669.0 (913.8) | 6285.8 (598.2)
  Cycle 1 Day 4 | 10837.5 (1299.4) | 7378.5 (770.8)
  Cycle 1 Day 8 | 5913.8 (614.8) | 4405.0 (639.8)
  Cycle 1 End | 2010.8 (187.7) | 1723.0 (127.9)
  10 min prior to initiation of Cycle 2 treatment | 1606.0 (169.8) | 1547.1 (196.82)
  Cycle 2 Day 3 | 7643.6 (1037.8) | 7017.7 (694.9)
  Cycle 2 Day 4 | 12439.5 (1670.7) | 11101.1 (1168.9)
  Cycle 2 Day 8 | 6481.0 (769.5) | 6124.0 (772.1)
  Cycle 2 End | 2065.9 (200.3) | 1931.7 (187.4)
  10 min prior to initiation of Cycle 3 | 2077.4 (188.6) | 1901.0 (214.3)
  Cycle 3 Day 3 | 9515.1 (1760.6) | 7636.7 (887.3)
  Cycle 3 Day 4 | 13907.1 (2319.7) | 13029.0 (1204.9)
  Cycle 3 Day 8 | 6705.8 (802.0) | 6879.2 (506.9)
  Cycle 3 End | 2334.8 (289.8) | 2198.8 (321.5)

9. Other Pre Specified Outcome: Tumor Vascularity
Time Frame: Up to 1 week
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Immunocytokine (IC) Binding
Time Frame: up to 1 week
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Interferon Gamma (INF-y) Expression
Time Frame: Up to 1 week
Reporting Status: Not Posted

12. Other Pre Specified Outcome: T Cell Reactivity
Time Frame: Up to 1 week
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Density of Cellular Infiltrate
Time Frame: Up to 1 week
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Expression of GD2 Target Antigen
Time Frame: Up to 1 week
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Natural Killer Cells (NK)
Description: NK and ADCC testing will be done on selected patients with freshly collected peripheral blood mononuclear cell (PBMC) at baseline (as a control), on day 8 of Courses 2 and 3, and on day 29/1 of Courses 2 and 3.
Time Frame: up to 12 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Antibody Dependent Cellular Cytotoxicity (ADCC)
Description: as for outcome 15
Time Frame: up to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 24 months
Description: Only Grade 3 and 4 Adverse Events (AEs) and AEs requiring dose modification are reported for this study.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 4/11 | 5/9 | 1/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/9 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 10/11 | 7/9 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=11) | Group B (N=9) | Group C (N=2) | Group D (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain - Head / Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=11) | Group B (N=9) | Group C (N=2) | Group D (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 10 (21) | 7 (18) | 2 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Tumor Pain
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seroma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic / Lab (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — AST
Metabolic / Lab (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — ALT/SGPT
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal Episode (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-01-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT00590824/Prot_SAP_000.pdf